CLINICAL TRIAL: NCT01115868
Title: An Exploratory, Single Centre, Randomized, Placebo Controlled, Assessor Blind Clinical Trial to Assess the Effects of Intradermal Administrations of Prevascar on Scarring in Human Subjects of African Continental Ancestral Origin
Brief Title: Prevascar in African Continental Group Scarring
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Renovo (Industry)
Responsible Party: Dr J Bush, Renovo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RN1003-0110
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2011-02

CONDITIONS: Scarring
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 2 - 2 doses of Prevascar and placebo (Experimental)
  Interventions: Drug: Prevascar 5ng; Drug: Prevascar 25ng; Drug: Prevascar 100ng; Drug: Prevascar 250ng
- Group 1 - 2 doses of Prevascar and placebo (Experimental)
  Interventions: Drug: Prevascar 5ng; Drug: Prevascar 25ng; Drug: Prevascar 100ng; Drug: Prevascar 250ng
- Group 3 - 2 doses of Prevascar and placebo (Experimental)
  Interventions: Drug: Prevascar 5ng; Drug: Prevascar 25ng; Drug: Prevascar 100ng; Drug: Prevascar 250ng
- Group 4 - 2 doses of Prevascar and placebo (Experimental)
  Interventions: Drug: Prevascar 5ng; Drug: Prevascar 25ng; Drug: Prevascar 100ng; Drug: Prevascar 250ng

INTERVENTIONS:
Drug: Prevascar 5ng — 100uL of 5ng/100uL Prevascar per linear centimetre wound margin injected intradermally.
Drug: Prevascar 25ng — • 100uL of 25ng/100uL Prevascar per linear centimetre wound margin injected intradermally.
Drug: Prevascar 100ng — • 100uL of 100ng/100uL Prevascar per linear centimetre wound margin injected intradermally.
Drug: Prevascar 250ng — • 100uL of 250ng/100uL Prevascar per linear centimetre wound margin injected intradermally.

SUMMARY:
There is considerable variation in scarring, within and between people, and between different ethnic groups. Individuals with more pigmented skin are more prone to severe scarring than those traditionally termed white. Prevascar is being developed by Renovo for use as a potential treatment for reducing scarring.

Renovo's histological analysis of wounds and scars in human non drug studies demonstrates an increase in wound and scar width in subjects of African Caribbean ancestry over a 12 month period.

It is hypothesised that IL-10 may be a potentially beneficial therapy for the reduction of scarring in Non Caucasians of African-Caribbean ancestry.

This Renovo clinical trial will be carried out primarily to establish the effects of four doses of Prevascar on 1cm incisional and excisional scars in subjects of African Continental Group ancestry, as compared to placebo, and to further investigate the safety and tolerance of intradermally injected Prevascar in wounds.

ELIGIBILITY:
Inclusion Criteria:

* Afro-Caribbean male and female subjects between 18 and 85 years of age.

Exclusion Criteria:

* Subjects who on direct questioning or examination have history or evidence of keloid scarring.
* Subjects who have evidence of any past or present clinically significant medical condition that would impair wound healing or trial assessments
* Subjects with a history of clinically significant hypersensitivity to any of the drugs or surgical dressings to be used in this trial.
* Subjects who are taking, or have taken, any investigational drugs within 3 months prior to the screening visit.
* Female subjects who are, or who become pregnant up to and including Day 0 and/ or who are lactating.
* In the opinion of the Investigator, a subject who is not likely to complete the trial for whatever reason.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-06 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
To assess the effects of Prevascar on resultant scars | 13 months
  To investigate the effects of Prevascar on wound/scar width
  To investigate the effects of Prevascar on wound/scar tissue histology
  To investigate the effects of Prevascar on scar appearance
  NB: This is an exploratory study and hence all objectives are exploratory

CONTACTS AND LOCATIONS:
Locations (1):
- Renovo Clinical Trials Unit, Manchester, Greater Manchester, United Kingdom